CLINICAL TRIAL: NCT02454725
Title: Regular HIV Testing Among At-Risk Latino Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO00020837; R34MH100947 (NIH)
Record Dates: First submitted 2015-04-20; First posted 2015-05-27 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: HIV Testing; Latino
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social Network (Experimental): Leaders of social networks will communicate messages endorsing regular HIV testing to network members.
  Interventions: Behavioral: Social Network; Behavioral: Comparison
- Comparison (Active Comparator): HIV counseling and testing
  Interventions: Behavioral: Comparison

INTERVENTIONS:
Behavioral: Social Network — Leaders of social networks will undergo small group training to develop skills to convey information effectively and deliver messages endorsing regular HIV testing to members of their social networks.
  Arms: Social Network
Behavioral: Comparison — All participants will receive HIV counseling and rapid testing following the Wisconsin Department of Health guidelines. Sexually active men who receive a negative test result will be told that they should be HIV-tested every three to six months, unless they have a monogamous HIV negative partner
  Other Names: HIV Counseling and Testing

SUMMARY:
Early HIV diagnosis followed by linkage to treatment soon after HIV infection can reduce mortality and prevent new HIV infections. To obtain the full benefit of early HIV diagnosis, the US Centers for Disease Control and Prevention suggest that high risk groups get tested for HIV regularly, every three to six months. This study will examine the feasibility of a strategy to promote regular HIV testing and HIV risk reduction among Latino men at risk for HIV which, if successful, will help to identify Latino men unaware of their HIV status, benefitting them and the society.

DETAILED DESCRIPTION:
In the US, the HIV epidemic largely affects clusters of interconnected persons with high HIV prevalence and undiagnosed HIV infections that must be reached to reduce incidence. Latino men who have sex with men (LMSM) are overrepresented in these clusters. Following African Americans, LMSM have the highest HIV incidence rate and are the next most likely to be unaware of their HIV infection. Between 2005 and 2008, nearly one-quarter of the HIV positive LMSM were unaware of the infection.

High HIV prevalence in LMSM networks and lack of strategies to promote regular HIV testing may explain why many LMSM are not benefiting from early diagnosis. Many LMSM face social and legal challenges that hinder their access to healthcare services and outreach. They often have little understanding of HIV treatments, experience discrimination, and hold mistaken assumptions about HIV risk, including beliefs that motivate them to seek sexual partners within their high prevalence in-group as a form of preventing infection.

A social network approach can address the demands of engaging LMSM in regular HIV screening and reduce their collective risk. LMSM often rely on other LMSM who are sources of advice and referrals and who partially shield them from the double jeopardy of being a sexual and ethnic minority. Network interventions can capitalize on these relationships to promote access to resources and foster norms that reward regular testing and encourage collective safety. This project uses social networks to promote regular HIV testing and risk reduction among LMSM. Rather than delivering risk reduction messages and opportunities for HIV testing, the intervention will penetrate networks of LMSM through well positioned members. Unlike strategies that target personal networks or social groups within venues, the intervention will recruit three-ring networks of interconnected LMSM and isolate their ties. Three recruitment rings will help to find less visible LMSM; and isolating their ties will identify who can reach them. In addition to informing and motivating their peers to reduce risk, key network members will be trained to be links to prevention resources, deliver tailored prompts to HIV testing, and support peers' testing behaviors to encourage repetition.

ELIGIBILITY:
Inclusion Criteria:

* self-report as a Latino man who has sex with men (LMSM);
* living in the Milwaukee area;
* willing and able to provide consent for participation;

Additional Inclusion Criteria for Social Network Seeds:

* more than 70% of social network members are LMSM
* more than 50% of LMSM social network members are at risk for HIV

Exclusion Criteria:

* Female
* 17 years of age or younger
* Unable to provide consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Frequency of HIV testing | Twelve months post intervention
  Maximum number of months between two HIV tests

SECONDARY OUTCOMES:
Frequency of HIV testing | Twelve months post intervention
  Whether the participant received an HIV test every < six months during the 12-month period following study intake
HIV risk behaviors: Number of unprotected anal intercourse occasions with a non-monogamous partner | Twelve months post intervention
  Number of unprotected anal intercourse occasions with a non-monogamous partner
HIV risk behaviors: Number of sexual partners | Twelve months post intervention
  Number of sexual partners

CONTACTS AND LOCATIONS:
Overall Officials: Laura R. Glasman, Ph.D., Principal Investigator — Medical College of Wisconsin